CLINICAL TRIAL: NCT01420159
Title: A Randomised, Double Blind, Multi-centre, Placebo Controlled Study to Evaluate the Efficacy and Safety of Methoxyflurane (Penthrox) for the Treatment of Acute Pain in Patients Presenting to an Emergency Department With Minor Trauma
Brief Title: Efficacy and Safety of Methoxyflurane (Penthrox) for the Treatment of Acute Pain in Minor Trauma
Acronym: STOP!
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Developments International Limited (Industry)
Collaborators: ORION Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEOF-001
Record Dates: First submitted 2011-08-11; First posted 2011-08-19 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Acute Pain Due to Trauma
Keywords: Pain; Trauma; Analgesia
MeSH Terms: conditions — Pain; Wounds and Injuries; Agnosia | interventions — Methoxyflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methoxyflurane (Experimental)
  Interventions: Drug: Methoxyflurane
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Patients will have access to two 3 mL methoxyflurane (Penthrox) Inhalers or two 5mL placebo Inhalers to be self-administered.
  Other Names: Penthrox

SUMMARY:
This study investigates the treatment of acute pain, an unpleasant feeling caused by an injury. The overall purpose of the study is to gain more information that the pain relief medicine Penthrox(Methoxyflurane) administered using the Penthrox Inhaler(a distinctive green, whistle like object that you breathe through) is safe and works at relieving pain in patients aged 12 years and older who are admitted to a hospital Emergency Department with a minor injury (known as trauma).

ELIGIBILITY:
Inclusion Criteria:

* Patients 12 years of age or older who are able to give written informed consent or who are accompanied by a parent(s)/legal guardian able to provide written informed consent on their behalf.
* Evidence of signed and dated informed consent document(s) indicating that the patient (and/or a parent/legal guardian) has been informed of all pertinent aspects of the study.
* Pain Score ≥ 4 to ≤ 7 as measured using Numerical Rating Scale (NRS) at the time of admission, due to minor trauma.

Exclusion Criteria:

* Life-threatening condition requiring immediate admission in the Operating Room or Intensive Care Unit.
* Presence of any other clinical condition(s) that may, in the opinion of the investigator, impact on the patient's ability to participate in the study, or on the study results, including history of head injury and/or altered consciousness.
* Unable to provide written informed consent.
* Known pregnancy or lactation
* Acute intoxication with drugs or alcohol, based on the judgement of the attending physician.
* Treatment with any analgesic agent within 5 hours prior to presentation to ED (except diclofenac sodium which is prohibited within 8 hours prior to presentation to ED).
* Current ongoing use of analgesics for chronic pain.
* Use of an investigational product within one month prior to presentation to ED.
* Known personal or familial hypersensitivity to fluorinated anaesthetics.
* Known personal or familial history of malignant hyperthermia.
* Clinically significant respiratory depression.
* Use of methoxyflurane in the previous 4 weeks.
* Known pre-existing clinically significant renal or hepatic impairment according to the judgement of the clinician.
* Clinically significant cardiovascular instability.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
VAS Score | Twenty Minutes
  The difference between treatment and placebo on the VAS pain score

SECONDARY OUTCOMES:
Rescue Medication | Up to a maximum of 6 hours
  A request for rescue medication, time of request for rescue medication and the quantity of opioid equivalent rescue medication administered will be measured
Time to pain relief | Up to a maximum of 6 hours
  The number of inhalations of study treatment until pain relief is achieved and the time until pain relief is achieved.
Responder analysis | Up to a maximum of 6 hours
  The number of responders will be defined
Safety Analysis | Up to 16 days
  Evaluation of Adverse Events experienced during treatment. Evaluation of Adverse Events, including safety laboratory samples, up to 14 +/- 2 days following Emergency Department discharge

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Coffey, Principal Investigator — Nottingham University Hospitals, Queen's Medical Centre Campus
Locations (6):
- United Kingdom (6):
  - Barnsley District General Hospital, Barnsley
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Colchester General Hospital, Colchester
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Queen's Medical Centre Campus, Nottingham

REFERENCES:
- [Derived] Hartshorn S, Dissmann P, Coffey F, Lomax M. Low-dose methoxyflurane analgesia in adolescent patients with moderate-to-severe trauma pain: a subgroup analysis of the STOP! study. J Pain Res. 2019 Feb 15;12:689-700. doi: 10.2147/JPR.S188675. eCollection 2019. PMID 30863141
- [Derived] Coffey F, Dissmann P, Mirza K, Lomax M. Methoxyflurane Analgesia in Adult Patients in the Emergency Department: A Subgroup Analysis of a Randomized, Double-blind, Placebo-controlled Study (STOP!). Adv Ther. 2016 Nov;33(11):2012-2031. doi: 10.1007/s12325-016-0405-7. Epub 2016 Aug 27. PMID 27567918
- [Derived] Coffey F, Wright J, Hartshorn S, Hunt P, Locker T, Mirza K, Dissmann P. STOP!: a randomised, double-blind, placebo-controlled study of the efficacy and safety of methoxyflurane for the treatment of acute pain. Emerg Med J. 2014 Aug;31(8):613-8. doi: 10.1136/emermed-2013-202909. Epub 2014 Apr 17. PMID 24743584